CLINICAL TRIAL: NCT03596099
Title: Rice Vinegar as an Intervention to Lower Blood Pressure in Adults With Prehypertension and 10-year CVD Risk <10%
Acronym: Rice-vinegar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mizkan Holdings Co., Ltd. (Industry)
Collaborators: ObvioHealth (Industry); Endothelix (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OBVIO_MIZ_001
Record Dates: First submitted 2018-07-06; First posted 2018-07-23 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Prehypertension
Keywords: Prehypertension; Rice vinegar; vinegar; acetic acid
MeSH Terms: conditions — Prehypertension | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm, parallel-group, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A unique randomization ID number will be assigned by ClaimIt to each enrolled subject and associated with the correct study product kit number; this number will be used throughout the study (includes study execution, safety reporting, compliance with the study product, and efficacy). Both the Mizkan rice vinegar active product (acetic acid) and placebo (no acetic acid) will be labeled identically and will be distinguishable only by the individual subject ID printed on the label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mizkan rice vinegar with acetic acid (Experimental): 200mL serving of a fruit-flavored beverage containing diluted Mizkan rice vinegar and 750mg acetic acid.
  Interventions: Dietary Supplement: Mizkan rice vinegar with acetic acid
- Mizkan rice vinegar without acetic acid (Placebo Comparator): 200mL serving of a fruit-flavored beverage containing diluted Mizkan rice vinegar that has undergone a freeze-drying process to remove the acetic acid
  Interventions: Dietary Supplement: Mizkan rice vinegar without acetic acid

INTERVENTIONS:
Dietary Supplement: Mizkan rice vinegar with acetic acid — 200mL serving of a fruit-flavored beverage containing diluted Mizkan rice vinegar and 750mg acetic acid.
  Arms: Mizkan rice vinegar with acetic acid
Dietary Supplement: Mizkan rice vinegar without acetic acid — 200mL serving of a fruit-flavored beverage containing diluted Mizkan rice vinegar that has undergone a freeze-drying process to remove the acetic acid
  Arms: Mizkan rice vinegar without acetic acid

SUMMARY:
This study is to assess the blood pressure lowering effect of rice vinegar when consumed over a 12-week period by healthy adults ages 30-65 years old with prehypertension. Study subjects will be recruited online via ClaimIt software platform and randomized to receive either the active rice vinegar-based drink or placebo and will visit the Endothelix research study site in Houston, Texas, 6 times during the study (Week -2, 0, 4, 8, 12 and 16). Here, subjects will undergo blood pressure monitoring, endothelial function, and laboratory assessments.

DETAILED DESCRIPTION:
Approximately 75 million American adults have hypertension with nearly one in every three adults experiencing a condition known as prehypertension (1). In 2013, more than 360,000 American deaths involved high blood pressure as a primary or co-morbid cause (2). In hypertensive patients, the probability of a first occurrence of heart attack and/or stroke is 70% and 80%, respectively (2). Dietary and lifestyle modifications may help some individuals maintain BP within normal ranges.

Studies of acetic acid, main component of vinegar, conducted with rat and human revealed mechanisms of potential blood pressure lowering (3-7). Also several human clinical trials to assess the efficacy of vinegar on blood pressure have previously been conducted in Japan. Kajimoto et al (2001, 2003) reported that continuous intake of 750 mg of acetic acid daily (approximately 15 mL of vinegar) reduces systolic blood pressure of adults with prehypertension as well as adults with hypertension (8-9). Sadou et al (2006) also reported similar effects with tomato vinegar in adults with prehypertension (750 mg daily acetic acid intake)(10).

The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC7) published by U.S. Department of Health and Human Services in 2003 defines prehypertension as blood pressure ranging from 120-139 mmHg systolic and 80-89 mmHg diastolic (11). JNC7 states that "prehypertension is not a disease category". Individuals with prehypertension are not candidates for drug therapy, rather they are recommended to practice lifestyle modification to reduce the risk of developing hypertension in the future. The Centers for Disease Control (CDC) shows the same position to JNC7 that a person who have SBP (120-139 mmHg) or DBP (80-89 mmHg) are prehypertension at risk stage (https://www.cdc.gov/bloodpressure/measure.htm). U S Food and Drug Administration (FDA) shows similar position in 21 C.F.R. § 101.74(a)(1) that "Hypertension, or high blood pressure, generally means a systolic blood pressure of greater than 140 millimeters of mercury (mm Hg) or a diastolic blood pressure of greater than 90 mm Hg. Normotension, or normal blood pressure, is a systolic blood pressure below 140 mm Hg and diastolic blood pressure below 90 mm Hg.". Recently issued guidance by the American College of Cardiology, the American Heart Association, and other collaborators (ACC/AHA) has emphasized the importance of 10-year CVD risk in categorization of blood pressure, which is calculated using an individual's systolic and diastolic blood pressure values, blood cholesterol levels, and medical history (12). The recommended treatment for an individual with a 10-year CVD risk <10% and blood pressure ≤139 mmHg systolic and ≤89 mmHg diastolic is lifestyle modification and not pharmacologic intervention. The target population for this study is not hypertension as defined by FDA and will align with the blood pressure category of "prehypertension" as defined by JNC7, recognized by CDC, and an additional inclusion criterion of a 10-year CVD risk <10% in recognition of the 2017 ACC/AHA report.

Its potential effects on blood pressure of acetic acid in humans with prehypertension (all clinical trials in Japan) provide a rationale for this evaluation with a Mizkan rice vinegar fruit drink containing 750 mg acetic acid. The purpose of this trial is to investigate the effect of vinegar delivering 750 mg acetic acid on blood pressure over a 12-week period in individuals with prehypertension and a <10% 10-year CVD risk. Additionally, the impact of 750 mg acetic acid as delivered in the vinegar drink on blood markers of the renin-angiotensin-aldosterone system and a marker of endothelial function will be assessed after 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Prehypertension (SBP 120-139mmHg and /or DBP 80-89mmHg)
* Males and females
* Must be between 30-65 years of age
* BMI: ≥18.5 kg/m2 and ≤34.9 kg/m2
* Stable body weight [self-reported weight gain or loss <5kg (11 lbs) in the past 3 months]
* Agree to comply with the study procedures
* Able to understand and sign the electronic informed consent
* Has reliable access to the internet and smartphone, and the necessary skills required to complete study tasks

Exclusion Criteria:

* SBP ≥140mmHg or SBP <120mmHg
* Use of tobacco, illegal drugs, or legal drugs known to impact blood pressure (BP), including but not limited to: amphetamine-type stimulants, cannabis, cocaine, heroin and other opioids, and MDMA
* Significant alcohol consumption (women: >3 drinks a day or >7 drinks a week; men: >4 drinks per day or >14 drinks per week)
* Women who are pregnant or nursing, and those planning to become pregnant
* Frequent heartburn, e.g., ≥2 days or more per week
* Use of anti-hypertensives, anti-depressants, immunosuppressants, drugs for hyperlipidemia, drugs that alter nutrient metabolism, and/or supplements targeting blood pressure reduction, and/or sustained use of NSAIDs within 30 days before randomization
* Regular use of polyphenol supplements and unwilling to stop use at the time of screening and for the duration of the study
* Self-identified as "high" consumer of vinegar-containing foods (e.g., 2 days or more per week consumption of a vinegar drink or significant volumes from such categories as salad dressings, pickled foods, etc.)
* History of chronic medical conditions, including but not limited to Type 1 or 2 diabetes, cardiovascular disease (including previous heart attack or stroke), kidney dysfunction (including chronic kidney disease), cancer
* An ASCVD 10-year risk score of ≥10% based on the ACC/AHA ASCVD calculator as performed by the Investigator or designee via the ASCVD Risk Estimator website (http://tools.acc.org//ASCVD-Risk-Estimator-Plus/#!/calculate/estimate/)
* Participation in a clinical research trial within 30 days prior to signing the eIC during screening
* Clinically significant findings from the laboratory assessments obtained during screening, as assessed by the Investigator or designee
* Allergy to any component of the vinegar or placebo products
* Unable to understand the study and undergo the informed consent process despite assistance
* Having more than one individual from a household participate in the study (to ensure prevention of mistaken consumption of incorrect investigational product)
* Investigator's discretion, e.g., subject deemed unsuitable or unreliable in follow-up to interaction with Investigator or site staff

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | Weeks 4, 8, 12, and 16
  To compare the change from baseline in systolic blood pressure at Weeks 4, 8, 12 (end of treatment), and 16 (end of study), in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.

SECONDARY OUTCOMES:
Changes in Diastolic Blood Pressure | Weeks 4, 8, 12, and 16
  To compare change from the baseline versus Weeks 4, 8, 12, and 16 in diastolic blood pressure in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.
Changes in Corresponding Blood Biomarkers | Week 12
  To compare the changes from baseline versus Week 12 in corresponding blood biomarkers (angiotensin II, aldosterone, renin activity, and ACE activity) in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.
Changes in Vascular Reactivity via VENDYS® | Weeks 4, 8, 12, and 16
  To compare changes from the baseline versus Weeks 4, 8, 12, and 16 in vascular reactivity to assess the endothelial function via VENDYS® measurements in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.

OTHER OUTCOMES:
Changes in Laboratory Values | Week 12
  To compare the changes from baseline versus Week 12 in CBC, sodium, potassium, chloride, creatine, eGFR, AST, ALT, GGT, bilirubin, glucose, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, hs-CRP, and oxidized LDL cholesterol), and urinalysis (single void sodium, creatinine) in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.
Assessment of Adverse Events | Week 12
  To assess adverse events at Week 12 in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.
Usability of the ClaimIt Software Platform | Week 12
  To assess usability of the ClaimIt software platform in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.
Changes in Body Weight and BMI | Weeks 4, 8, 12, and 16
  To assess changes from baseline in body weight and BMI (calculated from measured weight and height) will be compared at Weeks 4, 8, 12, and 16 in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks.
Changes in Dietary Intake | Week 12
  To compare the changes from baseline versus Week 12 in dietary intake in subjects with prehypertension who consume Mizkan rice vinegar active product (acetic acid) daily or placebo (no acetic acid) over a period of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Bazzano, MD, PhD, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - Primary Care Research Group, Atlanta, Georgia
  - Endothelix Research Site c/o Bellaire Cardiology Associates, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merai R, Siegel C, Rakotz M, Basch P, Wright J, Wong B; DHSc; Thorpe P. CDC Grand Rounds: A Public Health Approach to Detect and Control Hypertension. MMWR Morb Mortal Wkly Rep. 2016 Nov 18;65(45):1261-1264. doi: 10.15585/mmwr.mm6545a3. PMID 27855138
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Sakakibara S, Murakami R, Takahashi M, Fushimi T, Murohara T, Kishi M, Kajimoto Y, Kitakaze M, Kaga T. Vinegar intake enhances flow-mediated vasodilatation via upregulation of endothelial nitric oxide synthase activity. Biosci Biotechnol Biochem. 2010;74(5):1055-61. doi: 10.1271/bbb.90953. Epub 2010 May 7. PMID 20460711
- [Background] Na L, Chu X, Jiang S, Li C, Li G, He Y, Liu Y, Li Y, Sun C. Vinegar decreases blood pressure by down-regulating AT1R expression via the AMPK/PGC-1alpha/PPARgamma pathway in spontaneously hypertensive rats. Eur J Nutr. 2016 Apr;55(3):1245-53. doi: 10.1007/s00394-015-0937-7. Epub 2015 Oct 18. PMID 26476634
- [Background] Mitrou P, Petsiou E, Papakonstantinou E, Maratou E, Lambadiari V, Dimitriadis P, Spanoudi F, Raptis SA, Dimitriadis G. Vinegar Consumption Increases Insulin-Stimulated Glucose Uptake by the Forearm Muscle in Humans with Type 2 Diabetes. J Diabetes Res. 2015;2015:175204. doi: 10.1155/2015/175204. Epub 2015 May 6. PMID 26064976
- [Background] Honsho S, Sugiyama A, Takahara A, Satoh Y, Nakamura Y, Hashimoto K. A red wine vinegar beverage can inhibit the renin-angiotensin system: experimental evidence in vivo. Biol Pharm Bull. 2005 Jul;28(7):1208-10. doi: 10.1248/bpb.28.1208. PMID 15997099
- [Background] Kondo S, Tayama K, Tsukamoto Y, Ikeda K, Yamori Y. Antihypertensive effects of acetic acid and vinegar on spontaneously hypertensive rats. Biosci Biotechnol Biochem. 2001 Dec;65(12):2690-4. doi: 10.1271/bbb.65.2690. PMID 11826965
- [Background] (8) Kajimoto, O., et al. (2001). Effects of a drink containing vinegar on blood pressure in mildly and moderately hypertensive subjects. J Nutr Food, 2001, 4, 1-14
- [Background] (9) Kajimoto, O., Tayama, K., Hirata, H., Nishimura, A., Tsukamoto, Y. (2003). Hypotensive effects of drinks containing vinegar on high normal blood pressure and milk hypertensive subjects. J Nutr Food, 6(1), 51-68
- [Background] (10) Sadou et al. (2006). Antihypertensive Effect and Safety of a Drink ContainingTomato Vinegar in Case of Long-term Intake for Subjects with High-normal Blood Pressure or Mild Hypertension. Jpn Pharmacol Ther, 34, 6
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Carey RM, Whelton PK; 2017 ACC/AHA Hypertension Guideline Writing Committee. Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Synopsis of the 2017 American College of Cardiology/American Heart Association Hypertension Guideline. Ann Intern Med. 2018 Mar 6;168(5):351-358. doi: 10.7326/M17-3203. Epub 2018 Jan 23. PMID 29357392